CLINICAL TRIAL: NCT06138210
Title: The Effect of Exosomes Derived From Human Induced Pluripotent Stem Cell (GD-iExo-003) in Acute Ischemic Stroke: an Exploratory Study.
Brief Title: The Effect of GD-iExo-003 in Acute Ischemic Stroke
Acronym: ExoCURE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Guidon Pharmaceutics Ltd. (Industry)
Responsible Party: Principal Investigator, Junwei Hao, MD, Director of Neurology Department, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XMEC-2023-004
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
Keywords: exosome
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exosomes group (Experimental): Patients in this arm will be given exosomes derived from human induced pluripotent stem cell for injection once a day for 7 days.
  Interventions: Drug: exosomes derived from human induced pluripotent stem cell for injection
- Exosomes placebo group (Placebo Comparator): Patients in this arm will be given a placebo of exosomes derived from human induced pluripotent stem cell for injection once a day for 7 days.
  Interventions: Drug: a placebo of exosomes derived from human induced pluripotent stem cell for injection

INTERVENTIONS:
Drug: exosomes derived from human induced pluripotent stem cell for injection — Exosomes derived from human induced pluripotent stem cell for injection (3.0ml, 1×10^11particles/ml).
  Other Names: GD-iExo-003
  Arms: Exosomes group
Drug: a placebo of exosomes derived from human induced pluripotent stem cell for injection — Exosomes placebo, 3.0ml
  Other Names: GD-iExo-003 placebo
  Arms: Exosomes placebo group

SUMMARY:
This is a multicenter, randomized, double-blinded, placebo-controlled, dose-escalation trial. The objective of this study is evaluating safety and preliminary efficacy of intravenous exosomes derived from human induced pluripotent stem cell (GD-iExo-003) in acute ischemic stroke.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded, placebo-controlled, dose-escalation trial. This study will consist of 2 parts, with part 1 being a dose-escalation study and part 2 being an expanded safety study based on part 1 findings.

A traditional 3+3 dose escalation design will be implemented in part 1. Cohort 1: receive 2×10^9 particles/kg; cohort 2: 4×10^9 particles/kg and cohort 3: 8×10^9 particles/kg. If no dose-limiting toxicities (DLTs) are observed for 2 weeks after administration of the first injection, a new cohort will be enrolled at the next planned dose level. If DLTs are observed in 1 participant in the cohort, another 3 participants will be treated in the same dose level. Dose escalation will be stopped until DLTs are observed in >33% of the participants.

In part 2, 20 subjects will be randomized in a 1:1 ratio [exosome (n=10) or exosome placebo (n=10)]. The dose level will be determined by Data Safety Monitoring Board based on part 1.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke
* Age 18-70 years, inclusion of both genders
* Modified Rankin Scale score before stroke of 0-1
* NIHSS score 6-20 at inclusion that did not change by ≥4 points from screening to baseline assessment.
* Time of stroke onset is known and treatment can be started between day 1 and 7 of onset.
* Confirmation of hemispheric cortical infarct with magnetic resonance imaging or computed tomography
* Subjects who received intravenous thrombolysis or underwent mechanical reperfusion are eligible if they meet all other eligibility criteria.
* Adequate hepatic and renal function: serum aspartate aminotransferase ≤2.5× upper limit of normal; serum alanine aminotransferase ≤2.5× upper limit of normal; blood urea nitrogen ≤1.25× upper limit of normal; serum creatinine ≤1.25× upper limit of normal
* Adequate cardiac function.
* Subjects or legal representative can sign the informed consent and must be willing and able to comply with all aspects of treatment and follow-up schedule.

Exclusion Criteria:

* Presence of intracranial hemorrhage on CT including hemorrhagic stroke, epidural hematoma, subdural hematoma, intraventricular hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage or hemorrhagic transformation, etc.
* Presence of a lacunar or a brainstem infarct as the etiology of current symptoms.
* Evidence of brain tumor or history of epilepsy or traumatic brain injury.
* Subjects with present malignant disease.
* Subjects with severe comorbidities including immunodeficiency or coagulation disorders.
* Subjects with Alzheimer's disease, Parkinson's disease or other degenerative neurological disease.
* Ongoing systemic infection, severe local infection or taking immunosuppressants.
* Subjects with positive hepatitis B surface antibody (HBsAg) and positive hepatitis B core antibody (HBcAb), or HBsAg-positive virus carriers, positive hepatitis C antibody, positive syphilis antibody or HIV
* Allergy to the study products.
* Documented allergies
* Participation in any clinical trial in the last 3 months
* Inability or unwillingness to comply with the study schedule
* Pregnancy, childbearing potential (unless it is certain that pregnancy is not possible), oe breast feeding
* Other serious medical or psychiatric illness that is not adequately controlled
* Other circumstances that the investigator considers inappropriate for participation in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe adverse events | 90±7 days
  The proportion of patients who experienced severe adverse events.

SECONDARY OUTCOMES:
Favorable functional outcome | 90±7 days
  Rate of favorable functional outcome defined as a modified Rankin Scale (mRS, scores range from 0 to 6, with 0 to 2 indicating favorable outcome and 3 to 6 indicating unfavorable outcome including 6 as death) score of 0-2.
Functional outcome | 90±7 days
  The range of mRS scores by shift analysis.
NIHSS score change | 14±2 days
  The change of National Institutes of Health Stroke Scale (NIHSS) score of day 14 to baseline.
NIHSS score change | 90±7 days
  The change of National Institutes of Health Stroke Scale (NIHSS) score of day 7 to baseline.
Quality of Life (EQ-5D-5L) | 90±7 days
  The value of EQ-5D-5L score.
Barthel Index (BI) | 90±7 days
  The value of BI
MoCA | 90±7 days
  The value of MoCA

OTHER OUTCOMES:
Change of infarct volume | 14±2 days
  The infarct volume is measured by CT or MRI from the baseline to 14 days
Blood marker changes from baseline to discharge | at discharge, an average of 14 days
  A number of blood markers will be examined including C-reactive protein, glial fibrillary acidic protein, IL-1β, IL-6, IL-8, IL-10, Tumor Necrosis Factor-alpha.
Degree of cerebral edema changes from baseline to 48 hours | 48 hours
  Degree of cerebral edema changes from baseline to 48 hours.
Single-cell RNA sequencing of peripheral blood | 7±1 days
  Single-cell RNA sequencing of peripheral blood from baseline to day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, MD; PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data to other researchers.